CLINICAL TRIAL: NCT05333159
Title: Clinical Efficacy of SGLT-2 Inhibitor After Stent Implantation in Patients With Coronary Heart Disease and Diabetes Mellitus：a Prospective Cohort Study
Brief Title: The Efficacy of SGLT-2 Inhibitor in Patients With CAD and DM Undergoing PCI.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaofan Wu, MD, Beijing Anzhen Hospital
Other Study IDs: KS2022016
Record Dates: First submitted 2022-04-12; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Diabete Mellitus
Keywords: coronary artery disease; diabetes mellitus; percutaneous coronary intervention; SGLT-2 inhibitor; insulin resistance; platelet reactivity
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Insulin Resistance | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; Canagliflozin; empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Experimental: Subjects will be treated with SGLT-2 inhibitors (dapagliflozin, canagliflozin, empagliflozin) with or without conventional hypoglycemic drugs .
  Interventions: Drug: SGLT2 inhibitor
- Control: Subjects will be only treated with conventional hypoglycemic drugs.

INTERVENTIONS:
Drug: SGLT2 inhibitor — dapagliflozin 10mg once daily dose canagliflozin100mg once daily dose empagliflozin 0mg once daily dose
  Other Names: dapagliflozin; canagliflozin; empagliflozin
  Groups: Experimental

SUMMARY:
The study is to compare the effects of SGLT-2 inhibitors and other oral hypoglycemic agents in patients with coronary heart disease and diabetes mellitus undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
This is a single center, observational study designed to evaluate the efficacy of SGLT-2 inhibitors and other oral hypoglycemic agents in patients with coronary heart disease and diabetes mellitus who underwent percutaneous coronary intervention (PCI). 1424 subjects will be enrolled. All patients were divided into the SGLT-2 inhibitors group and other oral hypoglycemic agents group according to whether they were discharged with SGLT-2 inhibitors or not. The primary endpoint is adverse cardiovascular and cerebrovascular events (MACCE), composite of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke and unplanned coronary revascularization at 12 months after the index PCI. The key secondary endpoints are changes in insulin resistance index and platelet reactivity at 3 months and change in glucose and lipid metabolism at 12 months after the index PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with coronary heart disease and diabetes mellitus who underwent percutaneous coronary intervention.
3. Patients were provided informed consent before the procedure.

Exclusion Criteria:

1. History of diabetic ketoacidosis, type 1 diabetes, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy.
2. History of one or more severe hypoglycemic episode within 6 months before screening
3. Ongoing, inadequately controlled thyroid disorder.
4. History of hepatitis B surface antigen or hepatitis C antibody positive
5. Any history of or planned bariatric surgery.
6. Current use of a corticosteroid medication or immunosuppressive agent, or likely to require treatment with a corticosteroid medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease and diabetes mellitus who underwent percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 1424 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCEs) | 12 months
  MACCE, defined as a composite of cardiovascular death, non-fatal myocardial infarction, non-fatal myocardial stroke and unplanned coronary revascularization. Event rates are adjudicated by an endpoint committee based on the time to the first occurrence of MACCEs.

SECONDARY OUTCOMES:
Changes of insulin resistance index | 3 months
  Changes of insulin resistance index at baseline prior to drug administration and at 3 months after the index PCI.
Changes of platelet reactivity | 3 months
  Changes of platelet reactivity at baseline prior to drug administration and at 3 months after the index PCI.
Changes of fasting plasma glucose (FPG) level | 12 months
  Changes of FPG level at baseline prior to drug administration and at 3 months after the index PCI.
Changes of glycated hemoglobin (HbA1c) | 12 months
  Changes of HbA1c at baseline prior to drug administration and at 12 months after the index PCI.
Changes of plasma lipid parameters | 12 months
  Changes of plasma lipid parameters including triglycerides, high-density lipoprotein cholesterol and low density lipoprotein cholesterol and total cholesterol at baseline prior to drug administration and at 12 months after the index PCI.

CONTACTS AND LOCATIONS:
Overall Officials: xiaofan Wu, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No